CLINICAL TRIAL: NCT03917797
Title: Dose-response and Efficacy of Umbilical Cord-derived Mesenchymal Stromal Cells in Renal Systemic Lupus Erythematosus
Brief Title: Mesenchymal Stromal Cells (MSC´s) in Renal Lupus
Acronym: MSC-ROLE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de los Andes, Chile (Other)
Responsible Party: Principal Investigator, Fernando E. Figueroa MD, Program Director Translational Research in Cell Therapy, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Phase II Lupus MSC
Record Dates: First submitted 2019-04-02; First posted 2019-04-17 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Lupus Erythematosus, Systemic; Lupus Glomerulonephritis
Keywords: Systemic Lupus Erythematosus; Mesenchymal Stromal Cells; Lupus nephritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Superiority trial comparing MSCs versus Placebo in SLE patients with severe renal disease receiving Standard of Care treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking for patients, physicians providing patient care and outcome assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSC treatment (Experimental): Intervention: a previously selected dose of MSCs (Phase IIa) will be administered by i.v. infusion at baseline and 6 months of follow-up (total 12 months), to patients with Severe Renal SLE subject also to Standard of Care treatment with Methylprednisolone and Cyclophosphamide followed by Mycophenolate.
  Interventions: Biological: MSC treatment; Drug: Standard of Care
- Placebo (Placebo Comparator): Intervention: A Placebo (infusion vehicle) will be administered by i.v. infusion at baseline and 6 months of follow-up (total 12 months), to patients with Severe Renal SLE subject also to Standard of Care treatment with Methylprednisolone and Cyclophosphamide followed by Mycophenolate.
  Interventions: Drug: Standard of Care; Drug: Placebo

INTERVENTIONS:
Biological: MSC treatment — Umbilical cord-derived Mesenchymal Stromal Cell
  Other Names: Cellistem ® Lupus
  Arms: MSC treatment
Drug: Standard of Care — Methylprednisolone; Cyclophosphamide; Prednisone; Mycophenolate
  Other Names: Standard of Care for Lupus Nephritis
Drug: Placebo — MSC infusion vehicle
  Other Names: Placebo (for MSC)
  Arms: Placebo

SUMMARY:
Phase II Clinical Trial to Assess the dose-response and Efficacy of Umbilical Cord-derived Mesenchymal Stromal Cells (MSCs) in Severe Renal Systemic Lupus Erythematosus (SLE).

DETAILED DESCRIPTION:
Phase IIa trial of escalating doses of intravenous (i.v.) MSCs in active SLE, followed by a Phase IIb, triple blind, controlled assessment of the selected MSC dosing versus Placebo, in SLE patients receiving Standard of Care Therapy for Severe Renal Disease,

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling 1997 updated American College of Rheumatology (ACR) Criteria or 2012 SLICC Classification Criteria for SLE
* Seropositive for antinuclear (≥1:80) and/or anti-DNA antibodies
* Fulfilling following criteria for active renal disease:

Class III or IV proliferative disease (ISN/RPS) Renal Biopsy within 12 months plus...

Active Urinary Sediment (> 5 red blood cells/high-power field and/or >8 white blood cells/high-power field and/or cylindruria during the current flare).

UPC ratio ≥ 1

Exclusion Criteria:

* Estimated GFR < 40ml/min/m2
* Addition during prior 3 months of randomization of: Bolus methylprednisolone or new immunosuppressive drug or intravenous immunoglobulin (IVIG) or Plasmapheresis.
* Addition during prior 6 months of randomization of Cyclophosphamide
* Addition during prior 12 months of randomization of Biological anti-B cell therapy
* Coexisting uncontrolled morbidity; Pregnancy or planned Pregnancy within next 12 months; uncontrolled infection or neoplastic disease. Pending unresolved surgical indication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2019-04-02 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Achievement of Global Renal Response (GR) at Study Endpoint | 12 months
  Proportion of Patients that achieve Complete (CR) or Partial (PR) Renal Response at Endpoint

SECONDARY OUTCOMES:
Achievement of Complete Renal Response (CR) at Study Endpoint | 12 months
  Proportion of Patients that achieve CR criteria including: 1) Urinary Protein:Creatinine (UPC) ratio < 0.5; 2) estimated Glomerular Filtration Rate (GFR) ≥ 120 ml/min/m2, or at least 80% of baseline; 3) urinalysis < 10 red blood cells (RBC) and no RBC casts per high power field; 4) Prednisone dose ≤10 mg/day.
Achievement of Partial Renal Response (PR) at Study Endpoint | 12 months
  Proportion of Patients that achieve PR criteria including: 1) reduction of UPC ratio to at least 50% of baseline; 2) estimated GFR ≥120 ml/min/m2, or at least 80% of baseline; 3) Prednisone dose ≤10 mg/day.
Treatment Failure | 24 weeks and 12 months
  Proportion of Patients that fulfill any of the following criteria for Treatment Failure including: 1) Daily Prednisone dose cannot be reduced ≤ 10 mg at week 24; 2) Daily Prednisone is increased above 10 mg after week 24; 3) Introduction of a new immunosuppressive regimen, not included in the trial; 4) Use of Rituximab prior to month 12.
Response of SLE Responder Index (SRI). | 12 months
  Proportion of Patients that achieve SRI response, defined as a >4-point reduction in the SELENA-SLEDAI score, no new British Isles Lupus Assessment Group [BILAG] A organ domain score and no more than 1 new BILAG B score, with no worsening in physician's global assessment score versus baseline).
  The Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA) version of the SLE Disease Activity Index (SLEDAI) is employed for this calculation.(SELENA-SLEDAI score). The SELENA-SLEDAI score addresses 24 descriptors in 9 organ-systems. Disease worsening increases the score that ranges from 0-105.
  The BILAG addresses 97 items in organ-system domains, in an ordinal (A-E) scale, converted to a numerical (0-96) scale for usual calculations.
Selena Sledai | 12 months
  Average change in Selena Sledai Score in patients and controls
BILAG score | 12 months
  Average hange in BILAG score in patients and controls
Disease Flares | 12 months
  Proportion of patients that experience flares as defined in the Selena Flare Index (SFI). Mild/Moderate Flares are defined by change of 3 or more points in the SELENA-SLEDAI score. Severe Flares are defined as an increase in the SELENA-SLEDAI score to more than 12 points
Biomarker Response | 24 weeks and 12 months
  Changes in the levels of disease relevant biomarkers in peripheral blood/plasma, including 1) anti-dsDNA antibodies by ELISA; 2) complement proteins C3/C4 by nephelometry (mg/dL); 3) Percentage of CD4+ T helper cell subpopulations (Th1, Th17, Treg) and 4) B cell subpopulations (Naive, Memory, Transitional) by Flow cytometry; and 5) Cytokine Panel by Luminex, including Tumor Necrosis Factor (TNF) alpha, Transforming Growth Factor (TGF) Beta1, Interleukin (lL) 6, IL-17A, IL-10, B-cell activating factor/B Lymphocyte Stimulator (BAFF/BLys), Monocyte chemoattractant protein-1 (MCP-1/CCL2), C-X-C motif chemokine 10 (CXCL10), Interferon (IFN) gamma.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando F E, MD, Principal Investigator — Professor School of Medicine
Locations (2):
- Chile (2):
  - Clínica Universidad de los Andes, Santiago, Santiago Metropolitan
  - Hospital Barros Luco Trudeau, Santiago, Santiago Metropolitan